CLINICAL TRIAL: NCT03807219
Title: A Randomized, Multicenter, Prospective, Double-blind, Placebo-controlled, Clinical Trial in the Parallel Groups to Determine the Efficacy and Safety of a 60-day Use of the Magnox Comfort Compared to the Placebo in Subjects With NLC
Brief Title: The Study of Efficacy and Safety of a 60-day Use of the Magnox Comfort Compared to the Placebo in Subjects With NLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Naveh Pharma LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FS-MAG-1907
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Nocturnal Leg Cramps
Keywords: nocturnal legs cramps; legs cramps; NLC
MeSH Terms: conditions — Sleep-Wake Transition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnox Comfort (Active Comparator): 80 subjects will be on the Magnox Comfort arm.
  Interventions: Dietary Supplement: Magnox Comfort
- Placebo (Placebo Comparator): 80 subjects will be on the Placebo arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Magnox Comfort — Magnox Comfort (Magnesium (226 mg in equivalent), Vitamin E - 45 mg, Vitamin B6 - 2 mg.).
  Arms: Magnox Comfort
Other: Placebo — placebo
  Arms: Placebo

SUMMARY:
A randomized, multicenter, prospective, double-blind, placebo-controlled, clinical trial in the parallel groups to determine the efficacy and safety of a 60-day use of the dietary supplement Magnox Comfort compared to the placebo in subjects with nocturnal legs cramps

DETAILED DESCRIPTION:
At the beginning of the study, study subjects undergo a 14-day screening period during which the number of episodes of NLC is recorded. For further participation in the study, they must have at least 4 NLC episodes. Thereafter, an examination of compliance with the study requirements is performed and study subjects are randomized to one of the two groups: for a 60-day of IP use (1 capsule of Magnox Comfort daily) or to the control group (1 capsule of placebo daily).

ELIGIBILITY:
Inclusion Criteria:

1. The study subject is informed and he/she was given enough time to think on his participation in the study and signed the informed consent form before the beginning of any procedures;
2. A study subject is a man or a woman over the age of 45 years;
3. The study subject has an established diagnosis of the nocturnal legs cramps;
4. The study subject understands the Ukrainian language;
5. The study subject has satisfactory results of the neurological examination of both lower extremities;
6. The study subject has a telephone and can use it permanently;

Exclusion Criteria:

1. The onset of one of the non-inclusion criteria;
2. The study subject has less than 4 episodes of NLC during the 14-day screening period;
3. There is necessity for significant change in the treatment tactics.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
The number of episodes of NLC | The difference in count of nocturnal legs cramps documented in the trial, as compared between the study product and the placebo treated individuals, during a treatment period of 60-day.
  The study subject will record the number of episodes of nocturnal legs cramps in the study subject's diary

SECONDARY OUTCOMES:
Duration of NLC | The difference in duration of nocturnal legs cramps documented in the trial, as compared between the study product and the placebo treated individuals, during a treatment period of 60-day.
  The study subject will record the length of cramps in the diary
Severity of pain associated with NLC | The difference in severity of pain of nocturnal legs cramps documented in the trial, as compared between the study product and the placebo treated individuals, during a treatment period of 60-day.
  The study subject will record the severity of cramps in the diary using the visual analog scale from 0 to 10
Change in quality of life (SF-36) | The difference in quality of life documented in the trial, as compared between the study product and the placebo treated individuals, during a treatment period of 60-day.
  Study Short Form 36 Health Survey (SF-36) is one of the most widely used universal HRQoL scales, and it is widely used in the HRQoL measurement of general population, evaluation of clinical trials and health policy evaluation.
Changing in the sleep quality | The difference in sleep quality documented in the trial, as compared between the study product and the placebo treated individuals, during a treatment period of 60-day.
  The evaluation will be conducted using VAS (visual analog scale) from 0 to 5
Drop-out rate | The difference in drop-out rate documented in the trial, as compared between the study product and the placebo treated individuals, during a treatment period of 60-day.
  Counts of drop-out subjects

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Primor, Study Director — Naveh Pharma LTD
Locations (7):
- Ukraine (7):
  - Kharkiv City Clinic №9, Kharkiv, Kharkivs’ka Oblast’
  - Kyiv city clinic №9, Kyiv, Kyiv Oblast
  - Medical Center "Artem", Kyiv, Kyiv Oblast
  - Medical Center "Preventclinic" LLC, Kyiv, Kyiv Oblast
  - City clinic №5, Lviv, Lviv Oblast
  - Odesa Railway City Clinic, Odesa, Odesa Oblast
  - Medical center "Desna" LLC, Ternopil, Ternopil Oblast

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barna O, Lohoida P, Holovchenko Y, Bazylevych A, Velychko V, Hovbakh I, Bula L, Shechter M. A randomized, double-blind, placebo-controlled, multicenter study assessing the efficacy of magnesium oxide monohydrate in the treatment of nocturnal leg cramps. Nutr J. 2021 Oct 31;20(1):90. doi: 10.1186/s12937-021-00747-9. PMID 34719399